CLINICAL TRIAL: NCT00564018
Title: Duration of The Honeymoon Phase of Type 1 Diabetes: A Comparison of Insulins Detemir, Glargine and NPH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Presumed loss of clinical equipoise between the agents being investigated
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTSW-052006-056; 816 (Other: UT Southwestern Medical Center GCRC ID)
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes, basal-bolus, honeymoon, C-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Detemir (Experimental): 24 subjects randomized to therapy with a combination of insulins detemir and aspart at diagnosis of diabetes.
  Interventions: Drug: Insulin detemir
- Glargine (Experimental): 24 subjects randomized to therapy with a combination of insulins glargine and aspart at diagnosis of diabetes.
  Interventions: Drug: Glargine
- NPH (Experimental): 24 subjects randomized to therapy with a combination of insulins NPH and aspart at diagnosis of diabetes.
  Interventions: Drug: NPH

INTERVENTIONS:
Drug: Insulin detemir — Dosage adjusted to meet age-specific glycemic goals throughout course of study.
  Other Names: Levemir
  Arms: Detemir
Drug: Glargine — Dosage to be adjusted to meet age-specific glycemic goals throughout course of study.
  Other Names: Lantus
  Arms: Glargine
Drug: NPH — Dosage to be adjusted to meet age specific glycemic goals throughout course of study.
  Other Names: Neutral Protamine Hagedorn
  Arms: NPH

SUMMARY:
To determine whether using a long-acting insulin analog at the time of diagnosis, instead of intermediate-acting insulin, affects the rate of loss of the body's ability to make insulin in children with newly diagnosed type 1 diabetes.

DETAILED DESCRIPTION:
BACKGROUND: Type 1 diabetes (or insulin dependent diabetes mellitus (IDDM)) is a very common disorder affecting 1/400 persons by the age of 18 years and over 1 million people in the United States alone. An autoimmune disorder affecting the endocrine pancreas, it causes, in the untreated state, high blood glucose levels and ketosis. Over longer periods of time it can contribute to growth failure, malnutrition, and even death. It is responsible for a disproportionate percentage of the diabetes associated retinopathy and nephropathy seen in adults with diabetes (although type 1 diabetes only accounts for a small percentage of the total populace of patients with diabetes). Although insulin allows most children with this disease to grow and develop normally, it will not provide a permanent cure.

Many techniques have been studied to attempt to prevent the onset or progression of the autoimmune destruction of islets associated with type 1 diabetes, including a variety of immunomodulatory drugs, nicotinamide and small doses of insulin itself. Thus far nothing has proven completely successful. Some investigators have suggested that intensive control early in the disease process will slow the progression of the disease, but these results remain controversial. Ultimately, any treatment aimed at the prevention or cure of diabetes must have as its goal the preservation of the insulin secretory capacity of the pancreas.

In recent years, a number of insulin analogs have been developed which have different time-action profiles in humans. Currently, all children diagnosed with type 1 diabetes are placed on a combination of a long-acting insulin (such as insulins detemir or glargine) or a moderate-acting insulin (such as NPH), and a short acting insulin (such as lispro, aspart or regular insulin) as soon as they demonstrate they are able to resume a regular diet after their initial presentation. Each of the long- and moderate-acting insulins are given once or twice daily and the short-acting insulins at least twice and up to 4-5 times daily.

Normally, the pancreas secretes a basal level of insulin at rest, and then when challenged with a carbohydrate load, responds with an acute surge of insulin release. Intuitively, one might surmise that a pharmaceutical preparation that more closely mimics the normal physiological profile of the pancreas might be beneficial over the long term to pancreatic beta cell function. Levemir (insulin detemir) and Lantus (insulin glargine) are two relatively new insulin analogs known for their consistent and reproducible absorption profiles and steady time-action profiles. In comparison, insulin NPH is a product that had been the standard of care for children with diabetes for many years until the availability of the newer analogs, but is characterized by a peaking profile (with onset of action 2-4 hours after injection and peak effect 8-10 hours after injection). The combination of an insulin which mimics the basal insulin production of a pancreas at rest (i.e., glargine or detemir), together with a short-acting insulin with meals which mimics the bolus production of insulin generated in response to a carbohydrate load (regular, lispro or aspart), might allow for smoother blood glucose trends when compared to a combination of two "peaking" insulins (such as NPH and aspart).

In addition to the therapeutic benefit of better blood glucose control, we hypothesize that the maintenance of a steady baseline level of insulin with use of the newer insulin analogs may contribute to a longer period of pancreatic rest in the child newly diagnosed with diabetes. Many children with diabetes enter what is known as a "honeymoon phase" shortly after their diagnosis, which is characterized by relative ease of blood glucose control and relatively lower insulin requirements. This period represents a time during which the body is still able to make some insulin on its own.

We have retrospective data to suggest that children started on insulin glargine at diagnosis do, in fact, achieve significantly better glycemic control than age-matched children started on insulin NPH. This was assessed by HgbA1c measurements, which averaged a full percentage point lower at their 9 month visit for the glargine treated patients (Figure 1). A failure to see a significant improvement in patients switched from NPH to glargine well after diagnosis suggests that there is something to the initiation of treatment with glargine: perhaps the reason for improved control is a prolonged honeymoon period, in which the preservation of a small amount of innate insulin production allows for easier disease management.

What effect, if any, our current treatment modalities - specifically the choice of the longer acting insulin - have on the preservation of innate insulin secretory capacity remains unknown. If treatments aimed at the prevention or cure of diabetes are to maximize this secretory capacity, optimizing the insulin regimen may be imperative, and lack of attention to this parameter may confound trials of other interventions.

CONCISE SUMMARY OF PROJECT: Children aged 6-18 years who have been diagnosed with type 1 diabetes within the past 2 weeks will be randomized and placed in one of three treatment groups. 24 children will be randomized to each of three treatment arms differentiated by the choice of the longer-acting insulin (i.e. either detemir, glargine or NPH). All children will be treated with insulin aspart as the short-acting insulin to be used in combination with their longer-acting insulin. The insulin secretory capacity of the pancreas will be measured and compared between the groups by measuring C-peptide levels following a mixed meal tolerance test (using Boost) at 1, 6 and 12 months after diagnosis. Current standard of care as practiced at our institution is for these children to be seen every 3 months by a physician or advanced practice nurse at Children's Medical Center, Dallas. At each of these visits the children will have HgbA1c values measured and total daily insulin doses recorded. These will be secondary outcome measures for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 1 diabetes within 1 week of diagnosis
* Age 6 - 18 years
* Care provided at Children's Medical Center, Dallas

Exclusion Criteria:

* Actual treatment with oral drugs influencing beta cell function or blood glucose levels (e.g. oral hypoglycemic agents)
* Actual treatment with drugs influencing insulin sensitivity (e.g. Metformin, or systemic steroids)
* Significant concomitant disease likely to interfere with glucose metabolism (children with active bacterial infections at the time of diagnosis must be cured prior to entry)
* Expected poor compliance
* Pregnancy
* Any other condition that by the judgement of the investigator may be potentially harmful to the patients

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Adhikari, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Detemir: Subjects randomized to treatment with insulins detemir and aspart
- NPH Insulin: Subjects randomized to treatment with insulins NPH and aspart
- Glargine: Subjects randomized to treatment with insulins glargine and aspart
Period: Overall Study
Arm/Group | Detemir | NPH Insulin | Glargine
Started | 11 | 10 | 12
Completed | 9 | 7 | 11
Not Completed | 2 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who completed randomization into one of the three treatment arms
Groups:
- Isophane (NPH) Insulin: Subjects randomized to treatment with insulins NPH and aspart
- Total: Total of all reporting groups
Arm/Group | Detemir | Isophane (NPH) Insulin | Glargine | Total
Number analyzed (Participants) | 11 | 10 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects were recruited immediately after diagnosis of diabetes. Subjects who then tested (-) for type 1 diabetes associated antibodies were excluded from further analyses.
  years
    number analyzed (Participants) | 10 | 8 | 11 | 29
    (all) | 10.1 (3.0) | 11.0 (1.6) | 9.9 (2.5) | 10.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 9 | 19
  Male | 7 | 4 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 9 | 7 | 10 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 12 | 33
Hemoglobin A1c (percent) [Mean (Standard Deviation); unit: percent] — Population: Subjects were enrolled immediately after diagnosis of diabetes. Subjects who then were antibody (-) for type 1 diabetes associated antibodies are excluded from the baseline data reported.
  percent
    number analyzed (Participants) | 10 | 8 | 11 | 29
    (all) | 11.9 (1.7) | 12.6 (1.7) | 12.1 (1.8) | 12.2 (1.7)
Bicarbonate (HCO3) (meq/L) [Mean (Standard Deviation); unit: meQ/L] — Population: Subjects were recruited immediately after diagnosis of diabetes. Subjects who then tested (-) for type 1 diabetes associated antibodies were excluded from further analyses.
  meQ/L
    number analyzed (Participants) | 10 | 8 | 11 | 29
    (all) | 21.0 (4.7) | 15.6 (6.1) | 14.9 (8.1) | 17.3 (6.8)
Beta Hydroxy Butyrate (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — Population: Subjects were recruited immediately after diagnosis of diabetes. Subjects who then tested (-) for type 1 diabetes associated antibodies were excluded from further analyses.
  mmol/L
    number analyzed (Participants) | 10 | 8 | 11 | 29
    (all) | 4.7 (2.6) | 3.9 (3.5) | 7.9 (4.0) | 5.5 (3.6)
Total Daily Dose of Insulin (Units/kg/day) [Mean (Standard Deviation); unit: Units/kg/day] — Population: Subjects were recruited immediately after diagnosis of diabetes. Subjects who then tested (-) for type 1 diabetes associated antibodies were excluded from further analyses.
  Units/kg/day
    number analyzed (Participants) | 10 | 8 | 11 | 29
    (all) | 0.70 (0.11) | 0.69 (0.12) | 0.75 (0.14) | 0.70 (0.10)

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Area Under the Curve
Description: We measured the insulin secretory capacity of the pancreas by measuring C-peptide levels (and calculating the C-peptide area under the curve (AUC) using the trapezoidal method following a mixed meal tolerance test (using Boost) at 1, 6 and 12 months after diagnosis.
Time Frame: Although measured at 1, 6 and 12 months, the primary outcomes was a comparison between treatment groups at 6 months after diagnosis
Population: All subjects who completed 6 month mixed meal tolerance test (MMTT)s
Measure: Median (Inter-Quartile Range); unit: ng*hr/mL
Arm/Group | Detemir | NPH Insulin | Glargine
Number analyzed (Participants) | 10 | 7 | 10
ng*hr/mL | 220 [143 to 312] | 144 [83 to 302] | 51 [29 to 123]

2. Secondary Outcome: Glycemic Control as Determined by HgbA1c Values at 6 Months After Diagnosis
Description: We assessed glycemic control via measurement of Hemoglobin A1c at each quarterly clinic visit after diagnosis of diabetes. Data on the 6 month time point are presented
Time Frame: 6 months
Population: Data is presented for each subject at each time for which there was a measure.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Detemir | NPH Insulin | Glargine
Number analyzed (Participants) | 10 | 8 | 11
percent | 7.6 (1.3) | 8.0 (2.0) | 7.9 (1.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Detemir | NPH Insulin | Glargine
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12

LIMITATIONS AND CAVEATS:
Interpretation of the data is limited by the small sample sizes due to early study termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes